CLINICAL TRIAL: NCT07197957
Title: Clinical Utility of Cystatin C in the Early Detection of Contrast Induced Acute Kidney Injury
Brief Title: Cystatin and Early AKI Detection Contrast Induced Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: BayCare Health System (Other)
Responsible Party: Sponsor
Other Study IDs: Cystatin & Early AKI Detection
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the clinical utility of serum cystatin C in early detection of acute kidney injury (AKI).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the clinical utility of Cystatin C in early detection of contrast-induced AKI.

To evaluate the effect of patient characteristics in the Cystatin C based GFR estimation in comparison to Cr based estimation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18 years and above
* Inpatients with CKD (Figure 1)
* Order for CT imaging study or coronary angiography with isohexol Omnipaque) contrast media.
* Pre and post contrast available
* All races and ethnicity of patients are eligible. We expect to analyze approximately equal number of men and women in this study.

Exclusion Criteria:

* Preexisting dialysis
* Patients under the age of 18 years
* Pregnancy
* Incarcerated individuals
* Patients with impaired cognition and unable to follow consent procedures
* Recent exposure to CM (within 2 days before/after procedure)
* Cardiac shock
* Medications that affect biomarkers, including corticosteroids, lfamethoxazoletrimethoprim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be a cohort of inpatients with CKD. Eligible study participants, as defined by the inclusion criteria, will be consented at Morton Plant North Bay Hospital, Mease Countryside Hospital, and Morton Plant Hospital and St. Anthony's Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of AKI when sCr is used compared to when sCyC is used 24-48 hours after contract media and at 7-10 days follow-up | 10 days

SECONDARY OUTCOMES:
Change from baseline in eGFRcr compared to change from baseline in eGFRcys 24-48 hours after contrast media and at 7 to 10 days follow-up | 10 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Morton Plant Hospital, Clearwater, Florida
  - Morton Plant North Bay Hospital, New Port Richey, Florida
  - Mease Countryside Hospital, Safety Harbor, Florida
  - St. Anthony's Hospital, St. Petersburg, Florida